CLINICAL TRIAL: NCT02897401
Title: Determination of Carcinogens Nicotine in Electronic Cigarettes Users
Acronym: CANICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P150932
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Smoking; Carcinogenesis of the Nicotine
Keywords: urinary N'Nitrosonornicotine; nicotine; electronic cigarette; nicotine remplacement treatment
MeSH Terms: conditions — Smoking; Vaping | interventions — Pregnancy Tests; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Smocker (Experimental): Cigarette consumption in the context of their habit (not related to the particiapion under study).
  Interventions: Biological: pregnancy test; Biological: Urinary NNN assesement
- Electronic cigarette (Experimental): Electronic cigarette consumption in the context of their habit (not related to the particiapion under study).
  Interventions: Biological: pregnancy test; Biological: urinary cotinine assesment; Biological: Urinary NNN assesement; Behavioral: Questionnaire (Fagerstrom test); Procedure: Measurement of carbon monoxide levels expired
- Nicotine replacement therapy (Experimental): Nicotine replacement therapy (only patch) consumption in the context of their habit (not related to the particiapion under study).
  Interventions: Biological: pregnancy test; Biological: Urinary NNN assesement
- Without nicotine (Placebo Comparator): No consumption in the context of their habit (not related to the particiapion under study).
  Interventions: Biological: pregnancy test; Biological: urinary cotinine assesment; Biological: Urinary NNN assesement; Behavioral: Questionnaire (Fagerstrom test); Procedure: Measurement of carbon monoxide levels expired

INTERVENTIONS:
Biological: pregnancy test — Collection of 5 mL of urinary sample.The pregnancy test is done in each investigator center.
Biological: urinary cotinine assesment — Collection of 10 mL of urinary sample for cotinine analysis. The analysis is maid during the study and is centralised at the hospital Paul Brousse.
  Arms: Electronic cigarette; Without nicotine
Biological: Urinary NNN assesement — Collection of 20 mL of urinary sample for NNN analysis. The analysis is maid at the end of the study and is centralised in a laboratory located at Strasbourg.
Behavioral: Questionnaire (Fagerstrom test) — This questionnaire will permit to assess the smoking habits of the participants.
  Arms: Electronic cigarette; Without nicotine
Procedure: Measurement of carbon monoxide levels expired — This test will permit to determinate if the participant are axposed to passive smoking or not.
  Arms: Electronic cigarette; Without nicotine

SUMMARY:
Multicenter, national study, non-randomized , controlled, comparative with 4 independent groups (20 participants in each group). There are 3 experimental groups ("smocker", "nicotine replacement therapy" an "electronic cigarette") and 1 control group ("without nicotine").

The main objective of the study is to compare the level of urinary NNN in the electronic cigarette users versus the nicotine replacement therapy (patch) users.

DETAILED DESCRIPTION:
The study has only one visit taking place as below:

* Verification of inclusion and non-inclusion criteria.
* Collection of the informed consent of the subject Given the non-invasive nature of the procedure, a period of reflection will be given to the subjects, however, information and obtaining consent will be made during the same visit.
* Collection of 5 mL of required for the pregnancy test in women of childbearing age. This collection does not need to be fasting. If this test is positive, the subject will not be included in the study.
* Collection of 30 mL of urine needed for the cotinine and the NNN quantitative analysis.

This collection does not need to be fasting.

Then , the urine sample is divided into two vials stored at -80 ° C:

* a 10 mL vial for the cotinine analysis,
* a 20 mL vial for the NNN analysis.

  * Realization of the Fagerstrom test (FTCD) in order to evaluate subject smoking. This test is not done for the group 4 (group "without nicotine")
  * Measurement of carbon monoxide in exhaled air If after signing the consent, the subject realizes that he cannot urinate or he did not enough urine during the inclusion visiting, the subject can come back the next working day to make the urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Group1:

  * Adults (18 years old and more)
  * Exclusive daily smoker for more than 4 weeks, consuming 10 manufactured cigarettes per day or more
  * With health insurance
* Group 2:

  * Adults (18 years old and more)
  * Users of electronic cigarette EGO or MOD type for 4 weeks or more
  * Using a nicotine dosage of 12mg / ml or more for at least 4 weeks
  * Former smokers who consumed 10 cigarettes per day or more
  * Having completely stopped smoking for at least 4 weeks
  * No Subjected to passive smoking (verified by measuring carbon monoxide in exhaled air)
  * With health insurance
* Group 3:

  * Adults (18 years old and more)
  * People in patch 21 mg / 24h or 25mg / 16h in the fourth week or more treatment
  * Without taking oral nicotine or electronic cigarette for at least 4 weeks
  * Not subject to passive smoking (verified by measuring carbon monoxide in exhaled air)
  * Former smokers who consumed 10 cigarettes per day or more
  * Having completely stopped smoking for at least 4 weeks
  * With health insurance
* Group 4 (control group):

  * Adults (18 years old and more)
  * People Non-smoking, non-users of electronic cigarette, non-users of nicotine replacement therapy for at least 4 weeks
  * Not subject to passive smoking (verified by measuring carbon monoxide in exhaled air)
  * With health insurance

Patients in Groups 1, 2 and 3 must have a urinary cotinine ≥ 100 (ratio cotinine / creatinine - Determination Cotinine DRI). Patients in group 4 must have a urinary cotinine ≤ 10 (cotinine / creatinine ratio - Determination Cotinine DRI)

The thresholds of carbon monoxide from clinical experience are:

* Non current smoker: 0 to 5 parts per million (ppm)
* Passive smoker: 6 to 9 ppm
* Current active smoker : 10 ppm or more

Non inclusion criteria

* Rolling tobacco, cigars, cigarillos, pipe, bidi, chicha, cannabis smockers during the last 4 weeks
* Users tobacco snuff or chewing tobacco during the last 4 weeks
* Users of oral nicotine replacement therapy (gum, lozenges, inhalers, oral spray) during the last 4 weeks.
* Users of drug for smoking cessation aid other than nicotinic treatment: Varenicline, Bupropion, clonidine, Cytisine during the last 4 weeks
* Pregnant or breastfeeding women
* Non-compliant or unable to follow directions
* Refusing to sign the informed consent
* Refusing to do the urine collection
* Under guardianship or any other protective measures

Exclusion Criteria:

* Group 1, 2 and 3:

  -Having an urinary cotinine <100 (ratio cotinine / creatinine - Determination Cotinine DRI)
* Group 4 (control group):

  * Having an urinary cotinine> 10 (ratio cotinine / creatinine - Determination Cotinine DRI)

The determination of urinary cotinine levels will be carried out centrally. The result will not be available at the inclusion visit. The included patients who do not have the urinary cotinine levels required for their group, will secondarily excluded from the study.

The number of subjects in Groups 1, 2 and 3 with a ratio of cotinine would be less than 100 is expected to be negligible.A102

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
NNN urinary concentrations obtained in the group "electronic cigarette" versus group "nocotine replacement treatment". | At the inclusion
  The determination of urinary NNN of will be performed at the end of the study only for subjects with cotinine / creatinine ratio adequate.

SECONDARY OUTCOMES:
NNN urinary concentrations obtained in the group "electronic cigarette" versus group "smocker" | At the inclusion
  The determination of urinary NNN of will be performed at the end of the study only for subjects with cotinine / creatinine ratio adequate.
NNN urinary concentrations obtained in the group "electronic cigarette" versus group "no consumption of nicotine" | At the inclusion
  The determination of urinary NNN of will be performed at the end of the study only for subjects with cotinine / creatinine ratio adequate.
NNN urinary concentrations obtained in the group "nicotine replacement treatment" versus group "smocker" | At the inclusion
  The determination of urinary NNN of will be performed at the end of the study only for subjects with cotinine / creatinine ratio adequate.
NNN urinary concentrations obtained in the group "nicotine replacement treatment" versus "no consumption of nicotine" | At the inclusion
  The determination of urinary NNN of will be performed at the end of the study only for subjects with cotinine / creatinine ratio adequate.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dupont, MD, Principal Investigator — APHP, Paul Brousse Hospital
Locations (1):
- APHP, Paul Brousse Hospital, Villejuif, France

IPD SHARING:
Plan to Share IPD: No